CLINICAL TRIAL: NCT04993235
Title: Body Representation, Neuropsychological Profile and Socio-emotional Development in Children With Overgrowth Syndromes, With a Specific Focus on Functional Assessment of Patients With Beckwith-Wiedemann Syndrome and Sotos Syndrome
Brief Title: Body Perception and Representation in Overgrowth Syndromes, Behavioral Assessment and Neuropsychological Development
Acronym: Body-PROBAND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: University of Trieste (Other)
Responsible Party: Sponsor
Other Study IDs: RS2021_842
Record Dates: First submitted 2021-07-21; First posted 2021-08-06 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Sotos Syndrome; Beckwith-Wiedemann Syndrome; Overgrowth Syndrome; Body Image; Body Schema
Keywords: Neuropsychological profile; Behavioral assessment; Body perception; Body representation
MeSH Terms: conditions — Sotos Syndrome; Beckwith-Wiedemann Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Sotos Syndrome: Children and adolescents with Sotos Syndrome
  Interventions: Behavioral: NEPSY-II; Behavioral: CBCL and AQ questionnaires; Behavioral: BUT questionnaire and experimental tasks
- Beckwith-Wiedemann Syndrome: Children and adolescents with Beckwith-Wiedemann Syndrome
  Interventions: Behavioral: NEPSY-II; Behavioral: CBCL and AQ questionnaires; Behavioral: BUT questionnaire and experimental tasks
- Control group: Adolescents with typical development
  Interventions: Behavioral: BUT questionnaire and experimental tasks

INTERVENTIONS:
Behavioral: NEPSY-II — Participants with SS and BWS are administered with selected subtests assessing six different neuropsychological domains
  Groups: Beckwith-Wiedemann Syndrome; Sotos Syndrome
Behavioral: CBCL and AQ questionnaires — Parents of participants with SS and BWS are administered with questionnaires assessing behavioral problems and autistic traits
  Groups: Beckwith-Wiedemann Syndrome; Sotos Syndrome
Behavioral: BUT questionnaire and experimental tasks — A questionnaire, a computer-based task, a body-illusion paradigm and two psychophysical tasks assessing diverse levels of body perception and representation. These tasks are administered to adolescents of the three groups

SUMMARY:
Sotos Syndrome (SS) and Beckwith-Wiedemann Syndrome (BWS) are known as overgrowth syndromes as they involve an excessive growth of the whole body or of specific body parts. Beyond their primary physical problems, people with SS and BWS could present cognitive delay, socio-emotional and social behavior difficulties. For the SS, previous research reported impairments in specific neuropsychological domains and alterations of social behavior. Nevertheless, a description of the neuropsychological and behavioral profile in developmental age is still lacking. For the BWS, only in recent years alterations in social-cognitive development and in social behavior have started to gain attention of clinicians and researchers. However, no study has investigated the neuropsychological and behavioral functioning of children and adolescents with BWS. In this light, this research project aims at providing the first detailed description of the neuropsychological and behavioral profile of children and adolescents with SS and BWS.

Moreover, patients with SS and BWS experience structural alterations of their bodies and are early exposed to invasive diagnostical and medical procedures, which could interfere with the development of body representation. Body representation starts forming early in life through the integration of exteroceptive and interoceptive information, and plays a pivotal role in the social-cognitive development. Given the changes occurring in puberty and the crucial importance of body image in the relationship with peers, adolescence could be seen as a critical period for studying body representation. Thus, this project would investigate body representation at multiple levels (i.e. body image, body schema and interoceptive perception) and evaluate their impact on social-cognitive abilities in adolescents with SS and BWS. It is expected that both the clinical groups show alterations of body representation compared to healthy peers, and that these alterations could associate with impairments in affect recognition and regulation.

DETAILED DESCRIPTION:
Background and Rationale Sotos Syndrome (SS) and Beckwith-Wiedemann Syndrome (BWS) are known as overgrowth syndromes as they involve alterations in dimensions of the whole body or of specific body parts. SS is characterized by advanced bone age, macrocephaly, characteristic facies and cognitive delay. For the latter aspect, recent studies has described impairments in specific neuropsychological domains and alterations of social behavior. However, this evidence has been gathered in small and non-uniform samples, thus requiring further investigation. Moreover, a description of the neuropsychological and behavioral profile of SS in developmental age is still lacking. BWS is presented with macroglossia, exomphalos, lateralized overgrowth and hyperinsulinism as cardinal features, and is often associated with Wilms tumor and pathologies of internal organs. While the medical care of these primary issues has greatly improved, recently alterations in social-cognitive development and in social behavior have started to gain attention of clinicians and researchers. Nevertheless, no study has investigated the neuropsychological and behavioral functioning of children and adolescents with BWS.

Body representation is a complex, multi-faceted construct encompassing all the processes that allow to perceive, to experience and to be aware of our body. Body representation starts forming from the first months of life through the integration of exteroceptive and interoceptive information, and plays a crucial role in social-cognitive development. Children with SS and BWS experience structural alterations of their bodies and are early exposed to invasive diagnostical and medical procedures, which could interfere with the development of body representation. Given the changes occurring in puberty and the crucial importance of body image in the relationship with peers, adolescence could be seen as a critical period for body representation. Here, multiple levels of body representation (i.e., body image, body schema and interoceptive accuracy) are investigated in adolescents with SS and BWS compared to a control group of peers with typical development.

Aims The current study would provide a full description of the neuropsychological and behavioral profile of children and adolescents with SS and BWS (Aim 1). Moreover, this study protocol aims at investigating alterations of body representation at multiple levels, i.e. body image, body schema and interoceptive perception, and at evaluating their impact on social-cognitive abilities in adolescents with SS and BWS (Aim 2).

Methodologies This observational study involves two distinct assessment procedures, which may be conducted in a single session or in two sessions.

For Aim 1, children with SS and BWS are administered selected subtests of the NEPSY-II, the most adopted battery in developmental age in conditions of typical and atypical development. The NEPSY-II provides a full description of the neuropsychological profile in six different domains (Attention and executive functions, Language, Memory and learning, Sensorimotor functions, Social Perception, Visuospatial skills). Colored and Standard Raven's Matrices are also administered so as to obtain a reliable index of general intellectual functioning. Moreover, a standardized assessment of academic skills is performed by means of specific tests of the Memory and Transfert (MT) group for reading, comprehension and mathematic. Lastly, parents are asked to fulfil a sheet collecting socio-demographic and anamnestic information and two standardized questionnaires: the Child Behavior Check List (CBCL) assessing the presence of emotional-behavioral problems, and the Autistic Quotient (AQ) questionnaire assessing autistic traits related to five areas of functioning (social skills, attention switching, attention to detail, communication and imagination). The entire procedure is administered in a single session of approximately two hours and 30 minutes, in which short breaks between activities (approximately 10 minutes) are allowed so as not to overexert the child.

For Aim 2, adolescents (aged 11-18 years) with SS and BWS and healthy peers of the control group are administered with a self-report questionnaire assessing body image, an ad hoc created experimental task related to body schema, a virtual reality (VR) paradigm of full-body illusion and two psychophysical tasks assessing interoceptive accuracy. The Body Uneasiness Test (BUT) questionnaire consists of 34 items on a 1-5 Likert scale and allows for the assessment of five dimensions related to body image (weight phobia, body image preoccupation, compulsive self-monitoring, avoidance, and depersonalization). The experimental task, administered through a computer, was developed according to recent studies in literature that have assessed body schema changes in relation to peripersonal space and interpersonal distance. Specifically, participants observe inanimate objects or avatars approaching them. In one condition they have to judge whether they could easily reach the objects/avatars (peripersonal space), in the other condition they have to indicate when the object or avatar is perceived as "too close" (interpersonal distance). The full-body illusion paradigm involves the use of a camera placed 2 meters behind the participant and of a VR head mounted display. The back is touched by the experimenter and the image of this action is replayed to the participant synchronously or with a time delay, thus creating an incongruence between visual and haptic information.This paradigm induces an illusory sense of ownership of the virtual body to be elicited more effectively than tasks focused on individual body parts, and reliable as early as 7-8 year old. A short questionnaire adapted from the literature is administered after each condition so as to assess the illusion in terms of sense of ownership over the virtual body, sense of self location, and tactile sensations. In order to assess the ability to perceive interoceptive signals (interoceptive accuracy), participants are administerd a heartbeat perception task, in which they are asked to mentally count the number of their own heartbeats over a certain period of time. Their responses are compared with precise measurements of the heartbeats by means of a wrist-worn device that allows noninvasive determination of heartrate by photoplethysmography. The procedure is repeated in 4 different time intervals administered in random order among participants, without giving feedback on whether or not the responses are correct. In addition, a control task is proposed in which the participant are asked to mentally count the seconds elapsed in 3 time intervals. For both tasks, a visual analogic scale (VAS) is administered at the end of each time interval to assess the degree of confidence in providing the response (0 = totally unsure to 10 = extremely confident). Lastly, in order to assess the difference in heartrate perception at rest and in dynamic conditions, participants are administered the "Jumping Jack Paradigm," recently developed specifically for pediatric age (Schaan et al., 2019). For the baseline condition, participants, sitting in a comfortable position, are asked to indicate on a VAS how "loud" their heart rate feels. In the dynamic condition, participants are asked to jump for 10 s and then indicate again on VAS how loud they feel their heartbeat is. The responses provided on the VAS scales are compared with the heartrate recorded by the wrist-worn device. The physical activity required is minimal, thus posing no danger to participants. At the same time, this procedure facilitates the perception of the pulse and allows its assessment in an ecological and intuitive way, limiting the impact of any cognitive difficulties. The entire procedure is completed in approximately one hour and 30 minutes, inserting intervals of approximately 10 minutes between tasks.

Analysis Plan For the first aim, all variables will be transformed into scaled or standardized scores according to the normative tables for Italian samples, so as to compare performances of the clinical groups with the age-matched population with typical development.

For each clinical group, the neuropsychological and behavioral profile will be estimated using repeated-measures ANOVA models by entering the average scaled scores of each domain of the NEPSY-II and the standardized scores obtained in the behavioral scales of the CBCL questionnaire.

For the second aim, scores obtained in the five dimensions of the BUT questionnaire from the clinical groups will be compared to those of the control group by means of two-tailed Student's t-tests. For the body illusion task, the responses obtained at the questionnaire in the different conditions will be considered.

For the heartbeat perception task, the difference between actual and reported heartbeats will be transformed into an index of interoceptive accuracy according to previous literature. A similar measure will be estimated for the temporal accuracy control task by calculating the difference between actual and counted seconds.

For the experimental tasks, mixed ANOVA models will be used with both between-groups and within-subject factors (social/non-social stimulus for the computer-based behavioral task, synchronous and asynchronous stimulation for the full-body illusion, heart rate/seconds for the psychophysical tasks).

Significant interaction effects will be explored with post-hoc tests. For all analyses, the significance threshold will be set at p ≤ .05. Relationships between experimental task variables and those derived from standardized tests and questionnaires will be analyzed using Pearson's coefficient, correcting the significance threshold for the number of comparisons.

ELIGIBILITY:
Children and Adolescents with SS and BWS

Inclusion Criteria:

* diagnosis of Sotos Syndrome/Beckwith-Wiedemann Syndrome

Exclusion Criteria:

* severe motor and sensorial deficits that could interfere with tasks execution

Adolescents with typical development

Exclusion Criteria:

* any neurological or psychiatric conditions (e.g., learning disability, behavioral disorders etc.)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: For Aim 1 and 2 participants with SS and BWS aged 5-18 years will be recruited in collaboration with AIBWS and ASSI Gulliver, associations dedicated to families of patients with SS and BWS. For Aim 2, adolescents with typical development will be recruited in local schools.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological domains (Attention and Executive Functions, Language, Memory and Learning, Sensorimotor Functions, Social Perception; Visual-Spatial Functions) | At the recruitment - 1 session of 2/2.30 hours
  Mean scaled scores of each domain. Scaled scores range from 1 to 20, with mean = 10 and standard deviation (SD) = 3. Scores lower than 4 indicate specific difficulties.
Emotional-behavioral problems | At the recruitment - 1 session of 10 minutes
  Standardized scores at the the Child Behavior Check List. Standardized scores are reported with mean = 50 and SD = 10. Scores higher than 64 indicate possible problems, scores higher than 69 indicate clinical problems

SECONDARY OUTCOMES:
Body Uneasiness Test questionnaire | At the recruitment- 1 session of 15 minutes
  Mean scores obtained in the five dimensions of Body image. Higher scores indicate higher problems.
Peripersonal space and interpersonal distance | At the recruitment- 1 session of 20 minutes
  Peripersonal space and interpersonal distance in meters with social and non-social stimuli (avatar and objects) presented through the computer-based task
Full-body illusion | At the recruitment- 1 session of 30 minutes
  Scores at the VAS assessing sense of ownership overt the virtual body, sense of self-location and tactile sensations. Higher scores indicate higher sense of ownership, self-location and tactile sensations over the virtual body.
Heartbeat perception task and time estimation task | At the recruitment- 1 session of 15 minutes
  Difference between self-perceived and device-recorded heartbeats/seconds
Jumping Jack Paradigm | At the recruitment- 1 sessions of 10 minutes
  Difference between recorded heartbeats and scores at the VAS assessing perceived heartbeats at rest and after physical activity. Higher differences represent lower interoceptive accuracy

CONTACTS AND LOCATIONS:
Locations (1):
- Associazione La Nostra Famiglia - IRCCS Eugenio Medea, Bosisio Parini, Lombardy, Italy